CLINICAL TRIAL: NCT00104780
Title: A Phase II, Open Label, Multi-center Study of EP2101 Therapeutic Vaccine in Patients With Stage IIIB, Stage IV, or Recurrent Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Vaccine Therapy in Treating Patients With Stage IIIB, Stage IV, or Recurrent Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Epimmune (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000415721; EPIMMUNE-EP2101-201; MCMRC-0461
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2006-03

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — incomplete Freund's adjuvant

INTERVENTIONS:
Biological: EP-2101
Biological: incomplete Freund's adjuvant

SUMMARY:
RATIONALE: Vaccines made from peptides may make the body build an effective immune response to kill tumor cells.

PURPOSE: This phase II trial is studying how well vaccine therapy works in treating patients with stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with HLA-A2-positive, stage IIIB or IV or recurrent non-small cell lung cancer (NSCLC) treated with vaccine therapy comprising EP-2101 emulsified in montanide ISA-51 with that of historical controls and patients with HLA-A2-negative, stage IIIB or IV or recurrent NSCLC who undergo observation only.
* Determine the safety of this vaccine in these patients.

Secondary

* Determine progression-free survival of patients treated with this vaccine.
* Determine the frequency, magnitude, and breadth of cytotoxic and helper T-cell response to vaccine epitopes in patients treated with this vaccine.

OUTLINE: This is an open-label, multicenter study. Patients are assigned to 1 of 2 treatment groups according to HLA-A2 status.

* Group I (HLA-A2 positive): Patients receive vaccine therapy comprising EP-2101 emulsified in montanide ISA-51 subcutaneously once in weeks 0, 3, 6, 9, 12, and 15.
* Group II (HLA-A2 negative): Patients undergo observation in weeks 9 and 18. After completion of study treatment, patients in group I are followed at 3 weeks. All patients are then followed at months 1, 2, 3, 5, and 8, every 3 months for 2 years, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 84 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer meeting 1 of the following stage criteria:

  * Stage IIIB disease
  * Stage IV disease
  * Recurrent disease
* HLA-A2-positive disease

  * HLA-A2 negative patients are eligible to enroll in group II (observation) only
* Measurable disease
* Estimated tumor volume ≤ 125 cc
* No CNS signs or symptoms of brain metastases

  * Brain metastases that are clinically stable for ≥ 2 months AND do not require anticonvulsants or systemic steroids are allowed

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 12 weeks

Hematopoietic

* Hemoglobin ≥ 10 g/dL
* Platelet count > 100,000/mm^3
* WBC > 3,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Absolute lymphocyte count > 500/mm^3

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN for patients with liver involvement by tumor)
* Bilirubin ≤ 2.0 mg/dL (3.0 mg/dL for patients with liver involvement by tumor)
* Albumin ≥ 2.5 g/dL
* Alkaline phosphatase ≤ 2.5 times ULN
* No history of hepatitis B or C positivity

Renal

* Creatinine ≤ 2 times ULN

Immunologic

* No history of any of the following active conditions:

  * Systemic lupus erythematosus
  * Scleroderma
  * Connective tissue disease
  * Sjögren's syndrome
  * Multiple sclerosis
  * Rheumatoid arthritis
  * Inflammatory bowel disease
* No history of HIV positivity
* No history of serious adverse reaction, including anaphylaxis, or hypersensitivity to study vaccine or to any of its components

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 weeks after completion of study treatment
* No other malignancy within the past 5 years except curatively excised nonmelanoma skin cancer or surgically cured carcinoma in situ of the cervix
* No other acute medical condition that would preclude study treatment
* No mental or psychiatric condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 1 month since prior interferon therapy
* More than 1 month since prior interleukin therapy
* No prior cancer vaccine therapy, including participation in a vaccine study

Chemotherapy

* At least 4 weeks since prior chemotherapy

Endocrine therapy

* See Disease Characteristics
* More than 1 month since prior systemic corticosteroids except stable doses of inhaled corticosteroids

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* No concurrent participation in another investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12

PRIMARY OUTCOMES:
Comparison of overall survival with historical controls
Safety

SECONDARY OUTCOMES:
Progression-free survival
Frequency, magnitude, and breadth of cytotoxic and helper T-cell response to vaccine epitopes

CONTACTS AND LOCATIONS:
Overall Officials: Scott Plasman, Study Chair — Epimmune
Locations (9):
- United States (9):
  - Cancer Centers of Florida - Ocoee, Ocoee, Florida
  - New York Oncology Hematology, P. C. at Albany Regional Cancer Care, Albany, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Dayton Oncology & Hematology, P.A. - Kettering, Kettering, Ohio
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - Sarah Cannon Cancer Center at Centennial Medical Center, Nashville, Tennessee
  - Mary Crowley Medical Research Center at Sammons Cancer Center, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Cancer Care Northwest - North, Spokane, Washington